CLINICAL TRIAL: NCT04945863
Title: Association Between COVID-19 Vaccination and Reduced Mortality in Nursing Home Facilities.
Brief Title: COVID-19 in Nursing Homes 2020 and 2021
Status: Completed | Type: Observational
Sponsor: Lena Nilsson (Other)
Collaborators: Region Östergötland (Other)
Responsible Party: Sponsor-Investigator, Lena Nilsson, MD, Associate Professor, Chief Medical Officer, University Hospital, Linkoeping
Organization: University Hospital, Linkoeping (Other)
Other Study IDs: NH COVID 19
Record Dates: First submitted 2021-06-28; First posted 2021-06-30 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Comorbidities and Coexisting Conditions; Frailty; Covid19
MeSH Terms: conditions — Frailty; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To describe the effect on mortality in nursing home facilities during three separate equally long periods during the pandemic and more specifically to analyse the effect on mortality of improved preventive routines and vaccination.

DETAILED DESCRIPTION:
Retrospective descriptive cohort study in Östergötland County Council, Sweden comprising 136 nursing home facilities with a possibility to host 4500 residents. All residents in any of these NHs who had a laboratory confirmed COVID-19 diagnosis between March 2020 to April 2021 and who died within 30 days after the verified diagnosis are included. The study is undertaken as a retrospective record review. From the records patient-level data on demographic variables, clinical signs, comorbidity, performance status, and cause of death are collected.

ELIGIBILITY:
Inclusion Criteria:

* All residents in any of 136 nursing homes in Östergötland County Council, Sweden who had a laboratory confirmed COVID-19 diagnosis and who died within 30 days after the verified COVID-19 were included in three separate periods: First period from March 31 to June 30 2020; second period from October 15 2020 to January 15 2021; third period from January 16 to April 18 2021.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residents in nursing homes in Östergötland County Council, Sweden
Sampling Method: Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2021-04-18 (Actual); Study Completion 2021-04-18 (Actual)

PRIMARY OUTCOMES:
Comorbidity | March 2020 to April 2021
  Number of diagnoses bedisde COVID-19
Frailty | March 2020 to April 2021
  The combined assessment of performance status and frailty was adapted to the record review method
Cause of death | March 2020 to April 2021
  assessment of cause of death

CONTACTS AND LOCATIONS:
Locations (1):
- Anestesi- och operationskliniken, Universitetssjukhuset, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No